CLINICAL TRIAL: NCT05771103
Title: Stellate Ganglion Destruction With Alcohol Versus Thermal Ablation for Chronic Post Mastectomy Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AP2212-501-027
Record Dates: First submitted 2023-02-21; First posted 2023-03-16 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Post-mastectomy Pain Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stellate ganglion block with alcohol injection (Active Comparator): Stellate ganglion block with alcohol injection by ultrasound guidance and C7 level confirmation by fluoroscopy.
  Interventions: Device: thermal Radiofrequency neurolysis of Stellate ganglion
- thermal RF neurolysis of Stellate ganglion (Active Comparator): Stellate ganglion RF therapy will be done under fluoroscopy, integrated by ultrasound guidance
  Interventions: Device: thermal Radiofrequency neurolysis of Stellate ganglion

INTERVENTIONS:
Device: thermal Radiofrequency neurolysis of Stellate ganglion — Stellate ganglion block with alcohol injection versus thermal RF neurolysis of Stellate ganglion
  Other Names: Stellate ganglion block with alcohol injection

SUMMARY:
* Group A: SGB with alcohol injection by ultrasound guidance and C7 level confirmation by fluoroscopy.
* Group B: Thermal RF; thermal RF neurolysis will be applied with a time of 60 seconds at 80º C, and then will be repeated twice . Stellate ganglion RF therapy will be done under fluoroscopy, integrated by ultrasound guidance

DETAILED DESCRIPTION:
Breast cancer is the most common cause of cancer death for women . Postmastectomy pain syndrome (PMPS) is a frequent complication of breast surgery, and is considered a chronic neuropathic pain in the side of surgery which persists more than 3 months.

Complex regional pain syndrome (CRPS) is a clinical diagnosis with a highly variable presentation and prognosis. CRPS type I, previously known as reflex sympathetic dystrophy (RSD), is not associated with direct nerve injury. CRPS type II, or causalgia, is associated with direct injury of a specific nerve often from surgical intervention or trauma.

The stellate ganglion (SG), also known as the cervico-thoracic ganglion, is part of the sympathetic nervous system.

After assessment of eligibility criteria a predetermined randomization list and will be generated using random blocks.

* Group A: SGB with alcohol injection by ultrasound guidance and C7 level confirmation by fluoroscopy.
* Group B: Thermal RF; thermal RF neurolysis will be applied with a time of 60 seconds at 80º C, and then will be repeated twice has to be 0.5 cm apart from each other . Stellate ganglion RF therapy will be done under fluoroscopy, integrated by ultrasound guidance
* Group A ,The procedure will be started by placing the needle tip аntеrоlаteral to the lоngusсоlli muscle, dееp to the prеvеrtebrаlfаsсia in оrdеr tо аvоid spread along the carotid sheath, but superficial to the fascia investing the longus colli muscle (to prevent injecting into the muscle). Identifying the correct fascial plane achieved with portable ultrasound guidance thus facilitating the caudal spread of the injectate to reach the stellate ganglion at the C7-T1 level. This allowed for a more effective and stable sympathetic block with the use of a small injected volume. As an injection, we firstly used 1%-2.0 ml of lidocaine. The procedure will be continued by the injection of ethanol 50%, in quantity 1.5 ml for a lasting effect.
* Group B, thermal RF neurolysis will be applied with a time of 60 seconds at 80º C, and then will be repeated twice . Stellate ganglion RF therapy will be done under fluoroscopy, integrated by ultrasound guidance

ELIGIBILITY:
Inclusion Criteria:

* Female patient 20-65yrs underwent surgery for breast cancer
* Pain duration of more than 6 months
* Pain is moderate to severe pain (visual analog scale [VAS] ≥ 4 cm),
* Pain described as a refractory one that is defined as pain for which classic biomedical therapy has proven ineffective
* Pain is of positive neuropathic character as detected by the grading system for neuropathic pain (GSNP), with a score of 3 or 4

Exclusion Criteria:

* Refusal of the patient
* Recent myocardial infarction
* Anti-coagulated patients or coagulopathy (evaluate risk/benefit ratio)
* Glaucoma
* Pre-existing counter lateral nerve palsy
* Severe emphysema
* Cardiac conduction block
* Local and systemic sepsis
* Local anatomical distortion (which may render the block technically difficult or hazardous.
* Psychiatric illness.

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — female underwent radical mastectomy because of breast cancetr
Enrollment: 70 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Changes in VAS | 12 WEEKS
  assessment of pain relief pre and post neuro destruction of stellate ganglion 1, 4, 8 and 12 weeks . A 10 cm horizontal line version was used with 2 ends (left-end means no pain and right-end means the worst pain).
  Changes in VAS for assessment of pain relief pre and post neuro destruction of stellate ganglion 1, 4, 8 and 12 weeks. A 10 cm horizontal line version was used with 2 ends (left-end means no pain and right-end means the worst pain).
  Changes in VAS for assessment of pain relief pre and post neuro destruction of stellate ganglion 1, 4, 8 and 12 weeks. A 100 mm horizontal line version was used with 2 ends (left-end means no pain and right-end means the worst pain).

SECONDARY OUTCOMES:
patient satisfaction by patient satisfaction score and the analgesic concomitant medications consumption will be assessed before and 1,4,8 and 12 weeks after block | 12 weeks
  satisfaction score where 0 dissatisfied ,10 very satisfied

CONTACTS AND LOCATIONS:
Overall Officials: suzan adlan, lecturer, Principal Investigator — National Cancer Institute, Egypt
Locations (1):
- NCIEgypt IRB office, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No